CLINICAL TRIAL: NCT00151944
Title: A Phase III, Randomized, Multi-center, Open-label, 12 to 14 Month Extension Study to Evaluate the Safety and Tolerability of SPD476 (Mesalazine) Given Once Daily vs. Twice Daily for the Maintenance of Ulcerative Colitis in Remission.
Brief Title: Safety and Tolerability of SPD476 in Maintaining Remission in Patients With Ulcerative Colitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD476-303; 2004-000734-36 (EudraCT Number)
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

INTERVENTIONS:
Drug: SPD476 (mesalazine)

SUMMARY:
The purpose of this study is to test the long-term safety and tolerability of SPD476 in the maintenance of ulcerative colitis remission.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed all assessments of SPD476-301 or SPD476-302 End of Study/Early Withdrawal Visit
* Subjects who did not achieve remission at the End of Study/Early Withdrawal Visits in Study 301 or 302 will be eligible to enter the Acute Phase; subjects who did achieve remission at the End of Study Visits in Study 301 or 302 will be eligible to enter directly into the Maintenance Phase
* Women of childbearing potential must use an acceptable contraceptive method while on study treatment

Exclusion Criteria:

* Subjects who withdrew from Study 301 or 302 before Study Visit 3, or who withdrew due to a possible or probably related severe adverse event or serious adverse event are not eligible to enter this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-11-26 (Actual); Primary Completion 2006-03-13 (Actual); Study Completion 2006-03-13 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Throughout the study period of approximately 2 year, 4 months

SECONDARY OUTCOMES:
Time to relapse | Up to 12-14 months
Participant compliance | Up to 12-14 months
Number of participants in remission | 12 months
Ulcerative colitis disease activity index (UC-DAI) score | Baseline, Month 2, and Month 12
Patient questionnaire | Month 6, and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Result] Kamm MA, Lichtenstein GR, Sandborn WJ, Schreiber S, Lees K, Barrett K, Joseph R. Randomised trial of once- or twice-daily MMX mesalazine for maintenance of remission in ulcerative colitis. Gut. 2008 Jul;57(7):893-902. doi: 10.1136/gut.2007.138248. Epub 2008 Feb 13. PMID 18272546
- [Result] Kamm MA, Lichtenstein GR, Sandborn WJ, Schreiber S, Lees K, Barrett K, Joseph R. Effect of extended MMX mesalamine therapy for acute, mild-to-moderate ulcerative colitis. Inflamm Bowel Dis. 2009 Jan;15(1):1-8. doi: 10.1002/ibd.20580. PMID 18671232
- See also: FDA Recall information — http://www.fda.gov/opacom/7alerts.html
- See also: FDA-approved labelling information, US only — http://www.lialda.com/Professional/pdf/pi.pdf